CLINICAL TRIAL: NCT01027962
Title: Intensive Computerized Brain Training in Early Onset Psychosis-Pilot Phase
Brief Title: Intensive Computerized Brain Training (ICBT) in Youth With Early Onset Psychosis (EOP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Foundation of Hope, North Carolina (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Linmarie Sikich, MD, Associate Professor, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UNC # 09-0637; Maine #3589; R34MH085888-01 (NIH)
Record Dates: First submitted 2009-12-07; First posted 2009-12-09 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Psychosis
Keywords: Early Onset Psychosis; Laptop Computer; Brain Training
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ICBT Program (Other): Intensive Computerized Brain Training using software packages donated by Posit Science.
  Interventions: Other: ICBT Program
- Control Intervention (No Intervention): Commercially available computer games that do not contain violent stimuli but are appealing to youth between 10 and 19 years of age.
- Healthy Control Group (No Intervention): No participation in computer activity.

INTERVENTIONS:
Other: ICBT Program — Intensive Computerized Brain Training.
  Other Names: Posit Science
  Arms: ICBT Program

SUMMARY:
The purpose of this study is to examine whether an intensive computerized intervention targeted on improving central auditory and visual processing and executive functioning can be implemented in youths aged 10-19 with psychotic spectrum disorders, what developmental modifications are needed particularly for the younger participants, and whether it is possible to develop an appropriate, blinded control intervention.

DETAILED DESCRIPTION:
The purpose of this study is to provide a foundation for future rigorous study of an intervention that translates what we know about refinement of synaptic connections in response to environmental stimuli to an individualized intervention that directly improves neurocognitive functioning in youths with early onset psychosis(EOP). We will conduct a pilot randomized control study that determines the feasibility, tolerability and acceptability of Intensive Computerized Brain Training (ICBT) in youth with EOP.

Participants: Seventy youths, aged 10 years to 19 years inclusive will be assessed in the study. Forty youths with EOP will be randomly assigned to ICBT or an equally intense computerized game activity and 20 will be age, gender and race matched youths with no major psychiatric illnesses. We will allow for up to 5 EOP screen failures and up to 5 healthy control screen failures.

Procedures (methods): The forty participants with EOP will be randomly assigned to treatment with ICBT or equally intense video game play that also involves attention to sensory stimuli and requires increasingly skilled responses. A computer generated randomization schedule will be used to make assignments. Outcomes will be assessed at baseline, completion of the intervention (typically week 20), 3 after completing the intervention (typically month 8) and 7 months after completing the intervention(typically month 12). The other 20 youths, who comprise the typically developing comparison group known as healthy controls, will not participate in the computer activity or regular monthly psychiatric visits and will not complete satisfaction questionnaires. Up to 10 subjects may not be eligible to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

EOP participants:

* Clinical diagnosis of psychosis NOS, schizophrenia, schizoaffective, or schizophreniform disorder made by a child psychiatrist using DSM-IV criteria, confirmed by the KSADS (a semi-structured diagnostic interview) (Kaufman et al 1997)
* Age 10-19 years inclusive
* Guardian who is able and willing to participate in ongoing assessments and care
* Ongoing psychiatric care for EOP including medication treatment (except typical antipsychotic medication treatment)

Normal control participants:

* Age 10-19 years inclusive
* Guardian who is able and willing to participate in initial diagnostic assessment

Exclusion Criteria

EOP participants:

* Substance abuse within the month preceding treatment
* Hearing impairment that precludes participation in ICBT
* Visual impairment that precludes participation in ICBT
* Medical condition that is likely to impair learning or consciousness such as epilepsy or narcolepsy
* Lack of fluency in English language
* Severe psychotic symptoms that prevent quiet activity for up to 90 minutes at time
* Treatment with typical antipsychotic treatment
* Wide Range Achievement Test (WRAT (Wilkinson 1993)) word reading subscale grade equivalent of 2.9 or lower.
* Known history of premorbid developmental delay or learning disability
* Severe psychotic symptoms that prevent quiet activity for up to 90 minutes at time

Normal control participants:

* KSADS current or past diagnosis of psychiatric disorder including schizophrenia, schizoaffective disorder, schizophreniform disorder, psychosis NOS, bipolar disorder, major depression, obsessive compulsive disorder, panic disorder, post traumatic stress disorder, Tourette's disorder, eating disorder, borderline personality disorder, autism spectrum disorder, attention deficit disorder
* Family history in first or second degree relative of schizophrenia, schizoaffective disorder, schizophreniform disorder, psychosis NOS, bipolar disorder, major depression, substance abuse, obsessive compulsive disorder, panic disorder, post traumatic stress disorder, Tourette's disorder, eating disorder, borderline personality disorder, autism spectrum disorder
* Substance use within the month preceding treatment
* Psychotropic medication treatment
* Hearing impairment that precludes participation in ICBT
* Visual impairment that precludes participation in ICBT
* Medical condition that is likely to impair learning or consciousness such as epilepsy or narcolepsy
* Lack of fluency in English language
* Severe psychotic symptoms that prevent quiet activity for up to 90 minutes at time
* Wide Range Achievement Test (WRAT (Wilkinson 1993)) word reading subscale grade equivalent of 2.9 or lower.
* Known history of premorbid developmental delay or learning disability

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2009-10; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Feasibility, Tolerability and Acceptability of Intensive Computerized Brain Training (ICBT) in youth with EOP. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Lin Sikich, MD, Principal Investigator — University of North Carolina, Chapel Hill; Ann Maloney, MD, Principal Investigator — MaineHealth
Locations (1):
- University of North Carolina, Chapel Hill, Chapel Hill, North Carolina, United States